CLINICAL TRIAL: NCT04643899
Title: Evaluation of the Effects of Electrical Muscle Stimulation on Carbohydrate Homeostasis in Adult Patients With Obesity
Brief Title: Effects of Electrostimulation on Glycemic Control in Obesity
Acronym: ElectrOBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ildys (Other)
Collaborators: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILDYS-ISC2-2020001; ID-RCB (Other: 2020-A00484-35)
Record Dates: First submitted 2020-10-29; First posted 2020-11-25 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Obesity Adult Onset
Keywords: muscle electrostimulation; diabetes; endocrinology; physical activity; quality of life; obesity
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity; Obesity

STUDY DESIGN:
Intervention Model Description: * Monocentric; prospective; opened ; randomized; controlled study
  * Distribution of patients in groups according to a ratio (1: 1)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients benefiting only from the usual nutritional rehabilitation program G1a: diabetic patients G1b: non-diabetic patients
- Electrostimulation group (Experimental): Patients benefiting from the usual program AND muscle electrostimulation sessions G2a: diabetic patients G2b: non-diabetic patients
  Interventions: Device: Muscle Electrostimulation

INTERVENTIONS:
Device: Muscle Electrostimulation — * Scheduled sessions of 20 minutes per day; 5 days a week
  * In physiotherapy or in their room for the most dependent patients
  * Installation and monitoring by a physiotherapist or by the trained clinical research nurse
  * Modalities:
    * Device program n ° 1: 20mn (2mn of warm-up, 15mn of work at 75hz, then 3mn of recovery)
    * 4 electrodes (2 per thigh): large model (5 * 10 cm) for better comfort - Dura-Stick Plus model (reference 42200)
    * Gradual auto-increase of the intensity to the highest possible value tolerated, nevertheless allowing a contraction
  Other Names: Compex Pro Rehab ®; 253311x - REF 201010
  Arms: Electrostimulation group

SUMMARY:
This study evaluate the effects of muscle electrostimulation (MES) on carbohydrate homeostasis in adult patients with obesity. Its aims are also to evaluate the tolerance of feasibilty and the tolerance of MES and the impact on basal metabolism ; muscle mass (maintenance, gain or loss) in a context of calorie restriction ; physical capacities ; adherence to the usual rehabilitation program ; eating behavior : quality of life.

DETAILED DESCRIPTION:
Prevalence of adult obesity in general french population (≈15%) justifies the implementation of innovative care. Prescribing regular physical activity is one of the recommendations for managing obesity. However, patients find it difficult because of non-adapted offered activities; non-achievement concrete results despite the effort; difficulties to manage activities and to plan objective. Situation is seen as a failure and discourages patients. In addition, the obese patient may suffer from orthopedic disorders, cardiovascular contraindications, and the excessive weight in itself may force him to become sedentary. The recommendations on the practice of physical activity in the overall management of obesity are therefore not always applicable.

Muscle electrostimulation (MES) could therefore be an interesting additional tool in the management of obesity and particularly of glycemic control in obese patients suffering from type 2 diabetes.

Studies are still relatively few and present certain limits (small samples, short period of MES, very specific populations, few parameters evaluated, lack of consensus on the methods of MES, etc.). The results are nevertheless encouraging and call for the implementation of additional studies.

Investigators therefore propose a controlled, randomized, single-center study in a group of 60 adult patients suffering from severe or morbid obesity (BMI> = 35) in a 3-week rehabilitation stay.

The aims are to establish whether MES is a possible and interesting tool in the management of obesity, by checking the following hypotheses:

* control of carbohydrate metabolism is better when a MES is implemented;
* MES sessions improve patients' physical capacities and / or their tolerance to exercise;
* MES improves the quality of life of patients;
* MES improves patient adherence to the usual nutritional rehabilitation program;
* MES sessions are well tolerated and the accepted intensity nevertheless guarantees sufficient muscle stimulation.

ELIGIBILITY:
Inclusion Criteria:

* men and women over 18 years old and under 70 years old
* with severe or morbid obesity (BMI> = 35)
* with or without bariatric surgery
* able to understand and respect the protocol and its requirement
* who signed the consent prior to any other procedure protocol

Exclusion Criteria:

* major patients under guardianship / curatorship / legal protection
* pregnant patients
* patients with epilepsy
* with an implanted electronic/electrical device (cardiac pacemaker, intracardiac defibrillator, etc.)
* with a baclofen pump
* suffering from serious disorders of the arterial circulation in the lower limbs such as Peripheral Arterial Obstructive Disease (PAOD)
* suffering from abdominal or inguinal hernia
* suffering from cardiac arrhythmia
* suffering from skin lesions and/or infections foci on one or more areas where the electrodes are placed
* suffering from sensory disorders in the areas of stimulation
* patients unable to complete the entire program

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
Carbohydrate balance | Continuous measurement over the entire stay (Day 1 to Day 21)
  Evaluation of the time spent (%) above / in / below the patient's glycemic targets measured with a "Free Style" glycemic holter

SECONDARY OUTCOMES:
Homa Index | Change from baseline (Day 1) to week 3 (Day 21)
  Insulin resistance assessment
Quicki Index | Change from baseline (Day 1) to week 3 (Day 21)
  Insulin sensitivity assessment
Blood Glucose Levels | Continuous measurement over the entire stay (Day 1 to Day 21)
  Evaluation of the glucose levels (average, minimum, maximum)
Postprandial blood glucose | Continuous measurement over the entire stay (Day 1 to Day 21)
  Assessment of the number of postprandial hyper and hypoglycemia
Basal blood metabolism | Change from baseline (Day 2) to week 3 (Day 21)
  Blood chemistry analysis (lipid balance)
Impedance | Change from baseline (Day 2) to week 3 (Day 20)
  Bioelectrical impedance analysis of body composition
Maximal voluntary force | Change from baseline (Day 2) to week 3 (Day 21)
  Measurement of the maximum voluntary strength and endurance of the quadriceps
Six-minutes walk test (6MWT) | Change from baseline (Day 1) to week 3 (Day 20)
  Measurement of the distance traveled during the 6MWT
"Ricci & Gagnon" questionnaire | Change from baseline (Day 2) to week 3 (Day 21)
  Assessment of the level of physical activities and sedentary lifestyle
Adherence to the rehabilitation program | Evaluation at each sessions from Day 1 to Day 21
  Evaluation of the number of performed sessions compared to the expected for the proposed activities (collective balneotherapy, individual balneotherapy, supervised adapted physical activities, independent nordic walking) with analysis of the reasons for the differences
Anthropometry | Change from baseline (Day 1) to week 3 (Day 21)
  Weight (Kg) and height (cm) will be combined to report BMI in kg/m2
Quality of life, obesity and dietetics (QOLOD) rating scale | Change from baseline (Day 1) to week 3 (Day 21)
  Evaluation of quality of life - This scale gives 5 sub-scores ranging from 0 (worse outcome) to 100 (better outcome) for each explored dimension.
Visual analog pain scale | Evaluation at each sessions from Day 2 to Day 20
  Assessment of pain intensity during MES sessions with a visual analog scale
MES sessions check | Change from baseline (Day 1) to week 3 (Day 21)
  Record of session criteria (duration, program, maximum intensity, contraction Y/N)

CONTACTS AND LOCATIONS:
Overall Officials: Lena SEITE, MD, Principal Investigator — Fondation Ildys
Locations (1):
- CF Center - Fondation Ildys Site de Perharidy, Roscoff, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grosset JF, Crowe L, De Vito G, O'Shea D, Caulfield B. Comparative effect of a 1 h session of electrical muscle stimulation and walking activity on energy expenditure and substrate oxidation in obese subjects. Appl Physiol Nutr Metab. 2013 Jan;38(1):57-65. doi: 10.1139/apnm-2011-0367. Epub 2012 Nov 12. PMID 23368829
- [Background] van Buuren F, Horstkotte D, Mellwig KP, Frund A, Vlachojannis M, Bogunovic N, Dimitriadis Z, Vortherms J, Humphrey R, Niebauer J. Electrical Myostimulation (EMS) Improves Glucose Metabolism and Oxygen Uptake in Type 2 Diabetes Mellitus Patients--Results from the EMS Study. Diabetes Technol Ther. 2015 Jun;17(6):413-9. doi: 10.1089/dia.2014.0315. Epub 2015 Mar 3. PMID 25734937
- [Background] Joubert M, Metayer L, Prevost G, Morera J, Rod A, Cailleux A, Parienti JJ, Reznik Y. Neuromuscular electrostimulation and insulin sensitivity in patients with type 2 diabetes: the ELECTRODIAB pilot study. Acta Diabetol. 2015 Apr;52(2):285-91. doi: 10.1007/s00592-014-0636-5. Epub 2014 Aug 9. PMID 25107502
- [Background] Miyamoto T, Fukuda K, Kimura T, Matsubara Y, Tsuda K, Moritani T. Effect of percutaneous electrical muscle stimulation on postprandial hyperglycemia in type 2 diabetes. Diabetes Res Clin Pract. 2012 Jun;96(3):306-12. doi: 10.1016/j.diabres.2012.01.006. Epub 2012 Jan 30. PMID 22296854
- [Background] Vivodtzev I, Maffiuletti NA, Borel AL, Grangier A, Wuyam B, Tamisier R, Pepin JL. Acute Feasibility of Neuromuscular Electrical Stimulation in Severely Obese Patients with Obstructive Sleep Apnea Syndrome: A Pilot Study. Biomed Res Int. 2017;2017:3704380. doi: 10.1155/2017/3704380. Epub 2017 Jan 17. PMID 28194410